CLINICAL TRIAL: NCT01505582
Title: Inspiratory Muscle Training and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012_SBrumagne_IMT-LBP; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2012-01

CONDITIONS: Inspiratory Muscle Training; Low Back Pain; Respiratory Disorders
MeSH Terms: conditions — Low Back Pain; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle training (Experimental)
  Interventions: Other: Inspiratory muscle training
- Sham inspiratory muscle training (Sham Comparator)
  Interventions: Other: Sham inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Three times daily inspiratory muscle training (2x30 breaths) at an intensity of 60% Pi,max
  Other Names: Powerbreathe Classic
  Arms: Inspiratory muscle training
Other: Sham inspiratory muscle training — Three times daily inspiratory muscle training (2x30 breaths) at an intensity of 10% Pi,max
  Other Names: Powerbreathe Classic
  Arms: Sham inspiratory muscle training

SUMMARY:
Proprioceptive weighting changes may explain differences in postural control performance. In addition, the respiratory movement has a disturbing effect on postural balance. Postural balance seems to be impaired in individuals with respiratory disorders. Besides the essential role of respiration, the diaphragm may also play an important role in the control of the trunk and postural balance. Deficits in proprioception are found in a subgroup of patients with low back pain. In addition, disorders of respiration have been identified as strongly related to low back pain.

The aim of the study is to clarify whether inspiratory muscle training has a positive effect on proprioceptive postural control in individuals with recurrent low back pain.

ELIGIBILITY:
Inclusion Criteria individuals with low back pain:

* Age: 18-45 years old
* At least 1 year of low back pain with/without referred pain in buttock/thigh
* At least 3 episodes of disabling low back pain
* At least a score of 20% on the Oswestry Disability Index
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder, respiratory disease, pregnancy
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Smoking history

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proprioceptive postural control | 8 weeks
  Center of pressure displacement (force plate) in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven; Thierry Troosters, PhD, Principal Investigator — KU Leuven; Roeland Lysens, MD, PhD, Principal Investigator — KU Leuven; Peter Van Wambeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397